CLINICAL TRIAL: NCT02936024
Title: One Stage vs. Two Stage Gubernaculum Sparing Laparoscopic Orchidopexy: A Randomized Controlled Trial
Brief Title: One Stage vs. Two Stage Gubernaculum Sparing Laparoscopic Orchidopexy (GSLO)
Acronym: GSLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GSLO
Record Dates: First submitted 2016-10-07; First posted 2016-10-18 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cryptorchidism
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Two-Stage GSLO Technique (Experimental): Gubernaculum-sparing laparoscopic orchidopexy will be done in two stages
  Interventions: Procedure: Two-Stage GSLO Technique
- Control Group: One-Stage GSLO Technique (Other): Gubernaculum-sparing laparoscopic orchidopexy will be done in a single stage
  Interventions: Procedure: One-Stage GSLO Technique

INTERVENTIONS:
Procedure: Two-Stage GSLO Technique — The patient will initially receive the first stage of the two-stage technique which involves the ligation of testicular vessels laparoscopically, or transection of these vessels using cautery. After the first stage is complete, the patient will be seen approximately 3-6 months later for the second stage. The second stage of the procedure involves free mobilization of the testis and placement/fixation of the testicle in the scrotum.
  Arms: Intervention Group: Two-Stage GSLO Technique
Procedure: One-Stage GSLO Technique — The patient will receive only one surgical procedure during which ligation of testicular vessels is performed, as well as mobilization of the testis and placement/fixation of the testicle in the scrotum.
  Arms: Control Group: One-Stage GSLO Technique

SUMMARY:
Undescended Testis (UDT) is the most common congenital anomaly of the genitalia in boys and it is commonly managed by surgical intervention. Patients with intra-abdominal or non palpable testis, specifically, are often managed using a laparoscopic assisted orchidopexy, a common surgical technique to bring undescended testes down into the scrotum. Evidence in the medical literature to support the superiority of either one stage or two stage gubernaculum sparing laparoscopic orchidopexy (GSLO) is lacking. Due to this reason, this study focuses on the effects of one stage versus two stage GSLO on a patient important outcome: testicular atrophy.

DETAILED DESCRIPTION:
The principal research question to be addressed is: what is the feasibility of a randomized controlled trial to assess whether in boys, 1-5 years of age, diagnosed with intraabdominal UDT, two-stage GSLO results in fewer postoperative testicular atrophies when compared to single-stage GSLO? The results of this study will be used to assess the feasibility of a randomized controlled trial on this topic. If our protocol does not require significant modifications, then participants assessed in this pilot trial will be included as participants in the definitive multicenter trial.

To the best of our knowledge, the full-scale trial will be the first prospective, multicenter, randomized controlled trial to study the success rates of single-stage and two-stage GSLO. The results of the definitive multicenter trial will inform guidelines both locally and nationally, regarding the efficacy of staged techniques for orchidopexy. The results of this study will also inform and improve current care for children with IAT, as atrophy rates can be as high as 33% using the traditional laparoscopic approach.

Furthermore, if it is shown that a single stage approach is more efficacious than a two-stage approach, it will limit unnecessary exposure of young children to general anesthetic, which may be associated with an increased risk for learning disability or behavioral problems

The control group will receive single-stage GSLO procedure, while the intervention group will receive a two-stage GSLO technique. The first stage of the two-stage technique involves the ligation of testicular vessels laparoscopically, or transection of these vessels using cautery. Approximately 3-6 months following the completion of the first stage, the patient is seen again and the second stage of the procedure is performed. Access is obtained with a Hasson technique through an umbilical incision. Dissection begins laterally and proceeds along the superior margin of the internal inguinal ring (IIR), extending medially beyond the obliterated umbilical artery, while preserving a wide strip of peritoneum between the testis and the gubernaculum. Further dissection is then performed proximally, near the bifurcation of the iliac vessels, which allows free mobilization of this peritoneal triangle containing collateral blood supply to the testis. Next, a laparoscopic grasper is advanced through the IIR alongside the gubernaculum, and into the most dependent aspect of the scrotum. The distal gubernacular attachments and preserved cremasteric vessels, along with the testis, are pulled through the IIR with the assistance of a laparoscopic grasper, following the normal testicular descent route into the ipsilateral scrotum. Upon completion of dissection and descent, the testis is fixed to the scrotum in a sub-dartos pouch with a single 4-0 polydioxanone (PDS) stitch. If the patient is randomized to receive single-stage GSLO procedure, it is important to note that both the ligation of testicular vessels and the mobilization of the testis occur during the same operation.

ELIGIBILITY:
Inclusion Criteria:

* boys 1-5 years of age at presentation to Pediatric Urology Clinics
* patients diagnosed with intraabdominal UDT
* patients who require one- or two-stage repair performed by fellowship-trained Pediatric Urologists

Exclusion Criteria:

* patients who have undergone previous laparoscopic orchidopexy
* patients with palpable testes
* patients requiring orchiectomy

Ages: 1 Year to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Testicular Atrophy at 3 Months | 3 months postoperatively
  How many children have been diagnosed with testicular atrophy 3 months after the surgery has been performed.
Rate of Postoperative Testicular Atrophy at 12 Months | 12 months postoperatively
  How many children have been diagnosed with testicular atrophy 12 months after the surgery has been performed.
Recruitment Rate | Through study completion, an average of 2 years
  Will be calculated as the percentage of eligible participants enrolled
Frequency of protocol violations | Through study completion, an average of 2 years
  Will be calculated as the number of protocol violations that occurred during the pilot phase of this trial.
Frequency of adverse events | Through study completion, an average of 2 years
  Will be calculated as the number of documented adverse events during the pilot phase of this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Braga, M.D., Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No